CLINICAL TRIAL: NCT03145064
Title: A Phase 2, Single Arm, Multicenter, Open-label Study of Bruton's Tyrosine Kinase (BTK) Inhibitor BGB-3111 in Subjects With Relapsed/Refractory Non-GCB Type Diffuse Large B Cell Lymphoma
Brief Title: Study of BTK Inhibitor Zanubrutinib in Participants With Relapsed/Refractory Non-GCB Type Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BGB-3111-207; CTR20170091 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Relapsed/refractory non-GCB type
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Participants received zanubrutinib BID.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Administered at a dose of 160 mg BID orally.
  Other Names: BGB-3111; BRUKINSA

SUMMARY:
Screening (up to 28 days); daily treatment until disease progression, unacceptable toxicity or death, withdrawal of consent, lost to follow-up, or study termination from sponsor; treatment (up to 2 years), safety follow-up (30 days); survival follow-up until data cutoff for final analysis.

DETAILED DESCRIPTION:
This is a single-arm, multicenter, open-label Phase 2 study to evaluate efficacy, safety, tolerability of BGB-3111 (zanubrutinib) in participants with relapsed/refractory non-germinal center B-cell (GCB) type diffuse large B-cell lymphoma (DLBCL).

The study will enroll approximately 40 participants treated with zanubrutinib (160 milligrams [mg]) twice daily (BID). All participants in the study were treated until disease progression, unacceptable toxicity, death, withdrawal of consent, or the study was terminated by the sponsor for final analysis. At the time of final analysis, participants who remained on treatment were considered for participation in the extension study when eligible. A treatment cycle consisted of 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed non-germinal center DLBCL, by immunohistochemistry using the Hans algorithm:

   1. Cluster of differentiation 10 (CD10)- and B-cell lymphoma 6 protein (BCL6)-,
   2. CD10-, BCL6+, but maximal unique match+
2. Men and women ≥ 18 years of age.
3. Eastern Cooperative Oncology Group performance status of 0-2.
4. Measurable disease was defined as at least 1 lymph node > 1.5 centimeters in longest diameter and measurable in 2 perpendicular dimensions.
5. All participants must have provided fresh tumor biopsy or recent tumor tissue samples (within 2 years of study entry [informed consent form signed]).
6. Received at least one prior therapy for DLBCL that included anthracycline-based chemotherapy.
7. Participant not eligible for or refused intensive chemotherapy and hematopoietic stem cell transplant.
8. Documented failure to achieve at least partial response with, or documented disease progression after response to, the most recent treatment regimen.
9. Neutrophils ≥ 1 x 10^9/liter (L) independent of growth factor support within 7 days of study entry.
10. Platelets ≥ 75 x 10^9/L, independent of growth factor support or transfusion within 7 days of study entry.
11. Creatinine clearance of ≥ 30 milliliters/minute (as estimated by the Cockcroft-Gault equation or estimated glomerular filtration rate).
12. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN).
13. Bilirubin ≤ 2 x ULN (unless documented Gilbert's syndrome), then up to 5 x ULN allowed.
14. Independent of erythropoietin support or transfusion within 7 days of first dose of study drug.
15. International normalized ratio ≤ 1.5 and activated partial thromboplastin time ≤ 1.5 x ULN.
16. Participants may be enrolled who relapsed after autologous stem cell transplant if they are at least 6 months after transplant, participants should have had no active infections (that is, fungal or viral).
17. Females of childbearing potential must have agreed to use highly effective forms of birth control throughout the course of the study and at least up to 90 days after last dose of study drug. Highly effective forms of birth control were defined as abstinence, hysterectomy, bilateral oophorectomy with no menstrual bleeding for up to 6 months, intrauterine contraception, hormonal methods such as contraceptive injection, oral contraceptive. Males must have undergone sterilization-vasectomy, or utilized a barrier method where the female partner utilized the effective forms of birth control noted above.
18. Life expectancy of > 3 months.
19. Able to provide written informed consent and could understand and comply with the requirements of the study.

Key Exclusion Criteria:

1. Current or history of central nervous system lymphoma.
2. Prior exposure to a BTK inhibitor.
3. Prior corticosteroids (at dosages equivalent to prednisone > 20 mg/day) given with anti-neoplastic intent within 7 days, prior chemotherapy, targeted therapy, or radiation therapy within 3 weeks, or antibody-based therapies or Chinese anti-cancer herbal therapies within 4 weeks of the start of study drug.
4. Major surgery within 4 weeks of screening.
5. Toxicity of ≥ Grade 2 from prior anti-cancer therapy (except for alopecia, absolute neutrophil count [ANC]) and platelets. For ANC and platelets, please follow inclusion criteria #9 [neutrophils] and #10 [platelets]).
6. History of other active malignancies within 2 years of study entry, with exception of (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent.
7. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or history of myocardial infarction within 6 months of screening. Left ventricular ejection fraction is lower than 50% measured by echocardiography.
8. QTcF (Fridericia's correction) > 450 milliseconds or other significant electrocardiogram abnormalities including second degree atrioventricular (AV) block Type II, or third-degree AV block.
9. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
10. Uncontrolled systemic infection or infection requiring parenteral anti-microbial therapy.
11. Known human immunodeficiency virus, or active hepatitis B or hepatitis C infection (detected positive by polymerase chain reaction).
12. Pregnant or lactating women.
13. Any life-threatening illness, medical condition or organ system dysfunction, which, in the investigator's opinion, could compromise the participant's safety, or put the study at risk.
14. On medications that were strong cytochrome P450 (CYP), family 3, subfamily A (CYP3A) inhibitors or CYP3A inducers.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 41 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yang H, Xiang B, Song Y, Zhang H, Zhao W, Zou D, Lv F, Bai O, Liu A, Li C, Tan Z, Wang W, Gui H, Novotny W, Huang J, Li Y. Zanubrutinib monotherapy for patients with relapsed or refractory non-germinal center diffuse large B-cell lymphoma: results from a phase II, single-arm, multicenter, study. American Society of Clinical Oncology. 2020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers in China, all of which enrolled participants. The first participant was dosed on 30 June 2017. Since the primary and secondary objectives were met and the analysis was complete, the sponsor ended the study on 03 September 2020 (Last patient last visit). As of the final database lock (15 October 2020), 41 participants were enrolled and treated with zanubrutinib.
Groups:
- Zanubrutinib: Participants received 160 milligrams (mg) of zanubrutinib twice daily (BID).
Period: Overall Study
Arm/Group | Zanubrutinib
Started | 41
Received At Least 1 Dose of Study Drug | 41
Completed | 0
Not Completed | 41
Not completed — Death | 24
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 6
Not completed — Study ended by sponsor once primary/ secondary analysis was complete and participants discontinued | 4
Not completed — Other: Transferred to Long term Extension (LTE) study BGB-3111-LTE1 (NCT04170283) | 4

BASELINE CHARACTERISTICS:
Groups:
- Zanubrutinib: Participants received 160 mg of zanubrutinib BID.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 41
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Grade 0 : Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; Lower grades indicate better outcome.
  Participants
    Grade 0 | 10
    Grade 1 | 27
    Grade 2 | 4
Hepatitis B Core Antibody [Count of Participants; unit: Participants] — All positive participants were undetectable for hepatitis B virus DNA assessment.
  Participants
    Positive | 13
    Negative | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants achieving either a partial response (PR) or complete response (CR) as determined by investigator according to the 2014 modification of the International Working Group (IWG) in Non-Hodgkin's lymphoma (NHL) Criteria.
Time Frame: Up to approximately 23 months
Population: The Safety Analysis Set, which included all participants who received any dose of study drug, was the analysis set used for the efficacy and safety analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 41
percentage of participants | 29.3 [16.13 to 45.54]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from first dose of zanubrutinib until first documentation of progression (by IWG on NHL criteria) or death, whichever occurred first.
Time Frame: Up to 3 years and 2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 41
months | 2.8 [2.56 to 5.45]

3. Secondary Outcome: Duration Of Response
Description: Duration of response was defined as the time from the date that the response criteria were first met to the date that progressive disease was objectively documented or death, whichever occurred first. Duration of response was summarized for responders (with a best overall response of CR or PR) only.
Time Frame: Up to 3 years and 2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 12
months | 4.5 [2.14 to NA] — NA = Not estimable due to insufficient number of participants with events

4. Secondary Outcome: Time To Response
Description: Time to response was defined as the time from the first dose of zanubrutinib to the documentation of first response. Time to response was summarized for responders (with a best overall response of CR or PR) only.
Time Frame: Up to 3 years and 2 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 12
months | 2.83 [2.6 to 3.2]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A treatment-emergent adverse event was defined as an adverse event that had an onset date or a worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days following study drug discontinuation (Safety Follow-up Visit) or initiation of new anticancer therapy, whichever occurred first.
Time Frame: From the time of informed consent to 30 days after the last dose of study drug (approximately Up to 3 years and 2 months)
Population: The Safety Analysis Set included all participants who received any dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 41
Participants
  Participants with at least1 TEAE | 36
  Serious TEAE | 12
  TEAE leading to treatment discontinuation | 4

6. Other Pre Specified Outcome: Overall Survival
Description: Overall survival was defined as the time from first dose of zanubrutinib until death due to any cause.
Time Frame: Up to 3 years and 2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 41
months | 8.4 [4.8 to NA] — NA = Not estimable due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From the time of informed consent to 30 days after the last dose of study drug (approximately up to 3 years and 2 months).
Description: A treatment-emergent adverse event was defined as an adverse event that had an onset date or a worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days following study drug discontinuation (Safety Follow-up Visit) or initiation of new anticancer therapy, whichever occurred first.
Arm/Group | Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 24/41
Serious Adverse Events (participants affected / at risk) | 12/41
Other Adverse Events (participants affected / at risk) | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=41)
Pneumonia (Infections and infestations) | 3
Abdominal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Death (General disorders) | 2
Gait inability (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=41)
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 5
Blood creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Urinary tract infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 2
Influenza like illness (General disorders) | 2
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03145064/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03145064/SAP_001.pdf